CLINICAL TRIAL: NCT04266925
Title: Preventing Youth Soccer Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Schwebel, University Professor of Psychology & Associate Dean, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: X160720002
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Results first posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Injuries; Sports Injury; Sports Injuries in Children
Keywords: youth soccer injury
MeSH Terms: conditions — Wounds and Injuries; Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3 referees (Experimental): Three referees were present on the field during these youth soccer matches.
  Interventions: Behavioral: 3 referees present
- 1 referee (Active Comparator): One referee was present on the field during these youth soccer matches.
  Interventions: Other: 1 referee present

INTERVENTIONS:
Behavioral: 3 referees present — We compared player behavior with one versus three referees present on youth soccer fields during match play. The time between these two matches ranged from a few hours to several weeks.
  Arms: 3 referees
Other: 1 referee present — We compared player behavior with one versus three referees present on youth soccer fields during match play. The time between these two matches ranged from a few hours to several weeks.
  Arms: 1 referee

SUMMARY:
A study is proposed to test whether adding additional referees to youth soccer matches may reduce the risk of injury to the children playing soccer. Publicly-open youth soccer games will be randomly assigned to have either one or three referees and videotaped. The videotaped games will then be watched to record risk-taking behavior by players, referee decisions, and other factors relevant to potential injury.

ELIGIBILITY:
Inclusion Criteria:

* unit of measurement was youth soccer teams playing in Birmingham, Alabama area league

Exclusion Criteria:

* teams serving children under age 9 or over age 11

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2017-08-26 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Schwebel, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Youth Safety Lab, University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
Data will be shared with qualified experts upon request by email to study PI David Schwebel

REFERENCES:
- [Derived] Schwebel DC, Long DL, McClure LA. Injuries on the Youth Soccer (Football) Field: Do Additional Referees Reduce Risk? Randomized Crossover Trial. J Pediatr Psychol. 2020 Aug 1;45(7):759-766. doi: 10.1093/jpepsy/jsaa050. PMID 32651582

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 youth soccer teams were included this randomized crossover design. All completed both arms.
Groups:
- 3 Referees First: Three referees were present on the field first during these youth soccer matches.
  3 referees present: We compared player behavior with one versus three referees present on youth soccer fields during match play. The time between these two matches ranged from a few hours to several weeks.
- 1 Referee: One referee was present on the field first during these youth soccer matches.
  1 referee present: We compared player behavior with one versus three referees present on youth soccer fields during match play. The time between these two matches ranged from a few hours to several weeks.
Period: 1 Referee Game (~1 Hour)
Arm/Group | 3 Referees First | 1 Referee
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0
Period: 3 Referee Game (~1 Hour)
Arm/Group | 3 Referees First | 1 Referee
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: youth soccer teams
Groups:
- Total: Total of all reporting groups
Arm/Group | 3 Referees | 1 Referee | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 26 | 49
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 12 | 16 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Injuries During Soccer Matches
Description: average number of injury events requiring player to leave the field or be attended by an adult, across all games in study
Time Frame: baseline through one hour, which is beginning of the game until the end of the game, averaged across games
Population: youth soccer teams
Measure: Mean (Standard Deviation); unit: average number of injuries per game
Arm/Group | 3 Referees | 1 Referee
Number analyzed (Participants) | 49 | 49
average number of injuries per game | .4 (.7) | .4 (.7)

ADVERSE EVENTS:
Time Frame: full study period of about 10 weeks
Description: clinicaltrials.gov definition used
Arm/Group | 3 Referees | 1 Referee
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/25/NCT04266925/Prot_SAP_000.pdf